CLINICAL TRIAL: NCT05774288
Title: A Prospective, Multi-center, Randomized, Controlled Non-inferiority Clinical Trial to Evaluate the Safety and Efficacy of Cera™ Patent Foramen Ovale Occluders.
Brief Title: Safety and Efficacy of Cera™ Patent Foramen Ovale Occluders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB-CM01-P-275
Record Dates: First submitted 2023-02-26; First posted 2023-03-17 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Patent Foramen Ovale; Cryptogenic Stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomized controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cera™ patent foramen ovale occluders (Experimental): Patients with cryptogenic stroke complicated with patent foramen ovale will be implanted with the Cera™ patent foramen ovale occluders according to the INSTRUCTIONS for Use (IFU).
  Interventions: Device: Cera™ patent foramen ovale occluders
- Another patent foramen ovale occluders (Active Comparator): Patients with cryptogenic stroke complicated with patent foramen ovale will be implanted with the Another patent foramen ovale occluders according to the INSTRUCTIONS for Use (IFU).
  Interventions: Device: Another patent foramen ovale occluders

INTERVENTIONS:
Device: Cera™ patent foramen ovale occluders — Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with the Cera™ patent foramen ovale occluders according to the INSTRUCTIONS for Use (IFU).
  Arms: Cera™ patent foramen ovale occluders
Device: Another patent foramen ovale occluders — Patients who meet all the inclusion criteria and don't meet the exclusion criteria will be implanted with the Another patent foramen ovale occluders according to the INSTRUCTIONS for Use (IFU).
  Arms: Another patent foramen ovale occluders

SUMMARY:
To evaluate the performance of Cera™ patent foramen ovale occluders developed by Lifetech Scientific (Shenzhen) Co., LTD;

DETAILED DESCRIPTION:
The purpose of this prospective, multi-center, randomized, controlled non-inferiority clinical trial was to evaluate the safety and efficacy of Cera™ patent foramen ovale occluders developed by Lifetech Scientific (Shenzhen) Co., LTD for the treatment of cryptogenic stroke complicated with patent foramen ovale. The study required the implant to follow instructions strictly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-60 years;
2. Be able to understand the purpose of the experiment, voluntarily participate in the experiment and sign the informed consent;
3. Patent foramen ovale was confirmed by at least one of the following conditions exists:

   1. Patent foramen ovale was confirmed by Transthoracic echocardiography (TTE) or Transesophageal echocardiography (TEE);
   2. The presence of medium or large right-to-left shunt was confirmed by Right-heart acoustic contrast (cTTE or cTCD);
4. It meets the clinical status of patent foramen ovale plugging indication, and at least one of the following conditions exists:

   1. Cryptogenic stroke complicated with patent foramen ovale, combined with one or more clinical risk factors;
   2. Cryptogenic stroke complicated with patent foramen ovale, combined with one or more anatomical risk factors of patent foramen ovale;
   3. Cryptogenic stroke complicated with patent foramen ovale, with clear deep vein thrombosis or pulmonary embolism, and not suitable for anticoagulant therapy;
   4. Cryptogenic stroke complicated with patent foramen ovale, but still recurred with antiplatelet or anticoagulant therapy.

Exclusion Criteria:

1. Carotid atherosclerotic stenosis was determined by the investigator based on CT or vascular ultrasound (> 50%);
2. Large cerebral infarction occurred within 4 weeks (MR/CT or DWI image ASPECTS score <6 points or infarction volume ≥70 ml or infarction area > 1/3 middle cerebral artery blood supply area);
3. Patients with intracardiac thrombosis or tumor, intracardiac vegetations;
4. Acute myocardial infarction or unstable angina within 6 months;
5. Left ventricular aneurysm formation or left ventricular wall movement disorder;
6. Mitral/aortic disease: including mitral stenosis or severe mitral regurgitation of any cause, severe aortic stenosis or severe aortic regurgitation, mitral or aortic valve vegetations or prior valve replacement surgery;
7. Dilated cardiomyopathy, LVEF < 35%, or other severe heart failure;
8. Patients with right-to-left shunt due to other causes, including atrial septal defect or perforated diaphragm;
9. Atrial fibrillation/atrial flutter (chronic or intermittent);
10. Pregnant or planning to become pregnant during the trial;
11. Patients with active endocarditis or other untreated infections or other hemorrhagic diseases;
12. Pulmonary hypertension or patent foramen ovale was a special channel;
13. Liver and kidney function impairment (ALT or AST > 3 times the upper limit of normal value, serum creatinine (Cr) > 2 times the upper limit of normal value);
14. Uncontrolled hypertension (> 180/100 mmHg);
15. Contraindication of antiplatelet or anticoagulant therapy, such as severe bleeding within 3 months, obvious retinopathy, history of other intracranial bleeding, and obvious intracranial diseases;
16. Coronary heart disease, hypertension, diabetes and other vascular diseases that are poorly controlled by drugs or other means;
17. The investigator determined that the patient was not suitable for implantation of PFO occluder (for example, the diameter of the base of the atrial septal tumor ≥25mm and the size of the foramen ovale ≥5mm) or the patient has contraindications for implantation of PFO occluder;
18. Thrombosis exists at the location or route of implantation;
19. Malignant neoplasms or other diseases with a life expectancy of less than 2 years;
20. Patients who could not be followed up during the trial;
21. Participate in clinical trials of other drugs or medical devices within three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of effective occlusion | 180 days after surgery
  Effective occlusion was defined as: 180 days after the surgery, Transthoracic echocardiography (TTE) showed that the position and shape of the occluder were normal, and no horizontal atrial shunt was observed. Re-examination by Contrast transthoracic echocardiography (cTTE) showed no or only a small amount of right-to-left shunt, that is, no microvesicles or less than 10 microvesicles/frame in left heart cavity after Valsalva and resting state.

SECONDARY OUTCOMES:
Success rate of occluder implantation technology | 7 days after surgery
  The success of occluder implantation technology is defined as successful intraoperative implantation of occluder and immediate Echocardiography confirmed that the shape and position of the sealing device were appropriate, no new pericardial effusion or valve regurgitation was found, and the perioperative patients survived.
Success rate of surgical implantation of occlusion | 7 days after surgery
  Successful occluder implantation was defined as successful implantation of occluder and routine postoperative hospitalization that there were no serious adverse events related to surgery.
Success rate of complete occlusion | 180 days after surgery
  Complete occlusion was defined as the Transthoracic echocardiography (TTE) showing occlusion 180 days after surgery The position and shape of the apparatus were normal, and no horizontal atrial shunt was observed. The results of Contrast transthoracic echocardiography (cTTE) were reviewed there was no right-to-left shunt, that is, no microbubbles in the left heart cavity after Valsalva and resting state.
Success rate of effective occlusion | 360 days after surgery
  Success rate of effective occlusion was defined as: Transthoracic echocardiography (TTE) showed the position and shape of the occluder 360 days after the operation Normal condition, no horizontal atrial shunt; Reexamination by Contrast transthoracic echocardiography (cTTE) showed no or few results in other words, there were no microbubbles or less than 10 microbubbles in the left heart cavity after Valsalva and resting state.
Recurrence or incidence of cryptogenic stroke during follow-up | 360 days, 2 years, 3 years, 4 years, 5 years after surgery
  Cryptogenic stroke was defined as a new focal cerebral ischemia confirmed by neuroimaging (cranial MRI or CT), which was performed After extensive vascular, cardiac, and blood evaluation, non-atherosclerotic, cardiogenic, or arteriolar obliterators were identified Cerebral infarction caused by the diagnosis of exclusion.
All-cause mortality rate | 360 days, 2 years, 3 years, 4 years, 5 years after surgery
  All-cause death is defined as death from any cause during the follow-up period.
Incidence of new atrial fibrillation and atrial flutter during follow-up period | 360 days, 2 years, 3 years, 4 years, 5 years after surgery
  atrial fibrillation and atrial flutter
Incidence of device-related serious adverse events during follow-up (including device-related thrombosis, embolic stroke, and peripheral stroke) | 360 days, 2 years, 3 years, 4 years, 5 years after surgery
  Arterial embolism, Atrioventricular block III degree, heart abrasion, infective endocarditis, severe hemolytic anemia, etc.);
Incidence of device defects. | 360 days, 2 years, 3 years, 4 years, 5 years after surgery
  Device defects refer to unreasonable risks that may endanger human health and safety under normal use of medical devices in clinical trials, such as label errors, quality problems and failures.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, Doctor, Principal Investigator — Fuwai Yunnan Cardiovascular Hospital
Locations (14):
- China (14):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital ，CAMS&PUMC, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou people'Hospital, Meizhou, Guangdong
  - The Second XiangYa Hospital of Central South University, Changsha, Hunan
  - The Third XiangYa Hospital of Central South University, Changsha, Hunan
  - The First Hospital Of JiLin Universitv, Changchun, Jilin
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Qilu Hospitalof Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, Shandong
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No